CLINICAL TRIAL: NCT02141282
Title: A Phase 2 Open-Label Study of the Efficacy and Safety of ABT-199 (GDC-0199) in Chronic Lymphocytic Leukemia Subjects With Relapse or Refractory to B-Cell Receptor Signaling Pathway Inhibitor Therapy
Brief Title: A Phase 2 Open-Label Study of the Efficacy and Safety of ABT-199 (GDC-0199) in Chronic Lymphocytic Leukemia (CLL) Subjects With Relapse or Refractory to B-Cell Receptor Signaling Pathway Inhibitor Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Collaborators: Roche-Genentech (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M14-032
Expanded Access: NCT03123029 (Available)
Record Dates: First submitted 2014-05-12; First posted 2014-05-19 (Estimated); Results first posted 2022-12-19 (Actual); Last update posted 2022-12-19 (Actual); Status verified 2022-11

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: Oncology; Chronic Lymphocytic Leukemia; Cancer of the blood and bone marrow
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Neoplasms | interventions — venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- ABT-199 after ibrutinib therapy (Experimental): Participants with ibrutinib-resistant or refractory chronic lymphocytic leukemia (CLL) received venetoclax tablets once daily (QD) until disease progression or study drug discontinuation; median time on treatment was 593 days. The starting dose was 20 mg daily, increasing over a period of 5 weeks up to the daily dose of 400 mg.
  Interventions: Drug: Venetoclax
- ABT-199 after idelalisib therapy (Experimental): Participants with idelalisib-resistant or refractory chronic lymphocytic leukemia (CLL) received venetoclax tablets once daily (QD) until disease progression or study drug discontinuation; median time on treatment was 1023 days. The starting dose was 20 mg daily, increasing over a period of 5 weeks up to the daily dose of 400 mg.
  Interventions: Drug: Venetoclax
- ABT-199 after ibrutinib therapy: Expansion Cohort (Experimental): Participants with ibrutinib-resistant or refractory chronic lymphocytic leukemia (CLL) received venetoclax tablets once daily (QD) until disease progression or study drug discontinuation; median time on treatment was 622 days. The starting dose was 20 mg daily, increasing over a period of 5 weeks up to the daily dose of 400 mg. Participants enrolled into the Expansion Cohort with bulky disease at study entry who were non-responders or those who showed signs of clinical progression after completing the ramp up to 400 mg either by clinical disease assessment or by CT/MRI scan between Week 6 to Week 12 may have been permitted to escalate venetoclax to a daily dose of 600 mg.
  Interventions: Drug: Venetoclax
- ABT-199 after idelalisib therapy: Expansion Cohort (Experimental): Participants with idelalisib-resistant or refractory chronic lymphocytic leukemia (CLL) received venetoclax tablets once daily (QD) until disease progression or study drug discontinuation; median time on treatment was 1189 days. The starting dose was 20 mg daily, increasing over a period of 5 weeks up to the daily dose of 400 mg. Participants enrolled into the Expansion Cohort with bulky disease at study entry who were non-responders or those who showed signs of clinical progression after completing the ramp up to 400 mg either by clinical disease assessment or by CT/MRI scan between Week 6 to Week 12 may have been permitted to escalate venetoclax to a daily dose of 600 mg.
  Interventions: Drug: Venetoclax

INTERVENTIONS:
Drug: Venetoclax — Each dose of venetoclax was to be taken with approximately 240 mL of water within 30 minutes after the completion of breakfast or the participant's first meal of the day.
  Other Names: ABT-199; VENCLEXTA®

SUMMARY:
This was an open-label, non-randomized, multicenter, Phase 2 study evaluating the efficacy and safety of ABT-199 in 127 participants with relapsed or refractory chronic lymphocytic leukemia (CLL) after B-cell receptor signaling pathway inhibitors (BCR PI) treatment.

ELIGIBILITY:
Inclusion Criteria:

* Participant must have a diagnosis of chronic lymphocytic leukemia (CLL) that meets 2008 Modified International Workshop on Chronic Lymphocytic Leukemia National Cancer Institute-Working Group (IWCLL NCI-WG) criteria
* Participant has relapsed/refractory disease with an indication for treatment
* Participant has refractory disease or developed recurrence after therapy with a B-cell receptor pathway inhibitor (BCR PI)
* Participant must have an Eastern Cooperative Oncology Group performance score of ≤ 2
* Participant must have adequate bone marrow function at Screening
* Participant must have adequate coagulation profile, renal, and hepatic function, per laboratory reference range at Screening

Exclusion Criteria:

* Participant has undergone an allogeneic stem cell transplant within the past year
* Participant has developed Richter's transformation confirmed by biopsy
* Participant has active and uncontrolled autoimmune cytopenia
* Participant has malabsorption syndrome or other condition that precludes enteral route of administration
* Participant is human immunodeficiency virus (HIV) positive or has chronic hepatitis B or hepatitis C virus requiring treatment
* Participant has known contraindication or allergy to both xanthine oxidase inhibitors and rasburicase

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2014-09-10 (Actual); Primary Completion 2021-12-22 (Actual); Study Completion 2021-12-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (15):
- United States (15):
  - Moores Cancer Center at UC San Diego /ID# 128535, La Jolla, California
  - University of California, Los Angeles /ID# 127262, Los Angeles, California
  - Stanford University School of Med /ID# 126495, Stanford, California
  - Georgetown University Hospital /ID# 127261, Washington D.C., District of Columbia
  - Emory Midtown Infectious Disease Clinic /ID# 131249, Atlanta, Georgia
  - Northwestern University Feinberg School of Medicine /ID# 126497, Chicago, Illinois
  - Beth Israel Deaconess Medical Center /ID# 134509, Boston, Massachusetts
  - Dana-Farber Cancer Institute /ID# 126496, Boston, Massachusetts
  - Columbia Univ Medical Center /ID# 128536, New York, New York
  - New York Presbyterian Hospital Weill Cornell Medical Center /ID# 129648, New York, New York
  - Univ Rochester Med Ctr /ID# 130011, Rochester, New York
  - The Ohio State University /ID# 127263, Columbus, Ohio
  - University of Pennsylvania /ID# 126860, Philadelphia, Pennsylvania
  - University of Texas MD Anderson Cancer Center /ID# 126498, Houston, Texas
  - University of Utah /ID# 130813, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols, analyses plans, clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous independent scientific research, and will be provided following review and approval of a research proposal and statistical analysis plan and execution of a data sharing statement. Data requests can be submitted at any time after approval in the US and/or EU and a primary manuscript is accepted for publication. For more information on the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- [Derived] Roberts AW, Ma S, Kipps TJ, Coutre SE, Davids MS, Eichhorst B, Hallek M, Byrd JC, Humphrey K, Zhou L, Chyla B, Nielsen J, Potluri J, Kim SY, Verdugo M, Stilgenbauer S, Wierda WG, Seymour JF. Efficacy of venetoclax in relapsed chronic lymphocytic leukemia is influenced by disease and response variables. Blood. 2019 Jul 11;134(2):111-122. doi: 10.1182/blood.2018882555. Epub 2019 Apr 25. PMID 31023700
- [Derived] Coutre S, Choi M, Furman RR, Eradat H, Heffner L, Jones JA, Chyla B, Zhou L, Agarwal S, Waskiewicz T, Verdugo M, Humerickhouse RA, Potluri J, Wierda WG, Davids MS. Venetoclax for patients with chronic lymphocytic leukemia who progressed during or after idelalisib therapy. Blood. 2018 Apr 12;131(15):1704-1711. doi: 10.1182/blood-2017-06-788133. Epub 2018 Jan 5. PMID 29305552
- [Derived] Jones JA, Mato AR, Wierda WG, Davids MS, Choi M, Cheson BD, Furman RR, Lamanna N, Barr PM, Zhou L, Chyla B, Salem AH, Verdugo M, Humerickhouse RA, Potluri J, Coutre S, Woyach J, Byrd JC. Venetoclax for chronic lymphocytic leukaemia progressing after ibrutinib: an interim analysis of a multicentre, open-label, phase 2 trial. Lancet Oncol. 2018 Jan;19(1):65-75. doi: 10.1016/S1470-2045(17)30909-9. Epub 2017 Dec 12. PMID 29246803
- See also: clinical study report synopsis — https://www.abbvieclinicaltrials.com/study/?id=M14-032&Latitude=&Longitude=&LocationName=#additional-resources-section

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Safety population: all participants who received at least one dose of venetoclax
Period: Overall Study
Arm/Group | ABT-199 After Ibrutinib Therapy | ABT-199 After Idelalisib Therapy | ABT-199 After Ibrutinib Therapy: Expansion Cohort | ABT-199 After Idelalisib Therapy: Expansion Cohort
Started | 43 | 21 | 48 | 15
Completed | 0 | 0 | 0 | 0
Not Completed | 43 | 21 | 48 | 15
Not completed — Adverse event, not related to progression | 8 | 1 | 3 | 1
Not completed — Adverse event, related to progression | 1 | 0 | 2 | 0
Not completed — COVID-19 infection | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 4 | 2
Not completed — Other, not specified | 14 | 11 | 23 | 9
Not completed — Progressive disease, Richter's | 4 | 1 | 1 | 1
Not completed — Progressive disease per protocol | 12 | 7 | 9 | 2
Not completed — Stem cell transplant | 1 | 0 | 1 | 0
Not completed — Study terminated by Sponsor | 0 | 1 | 0 | 0
Not completed — Subject non-compliance | 0 | 0 | 1 | 0
Not completed — Withdrew consent | 2 | 0 | 4 | 0

BASELINE CHARACTERISTICS:
Population: All treated participants
Groups:
- Total: Total of all reporting groups
Arm/Group | ABT-199 After Ibrutinib Therapy | ABT-199 After Idelalisib Therapy | ABT-199 After Ibrutinib Therapy: Expansion Cohort | ABT-199 After Idelalisib Therapy: Expansion Cohort | Total
Number analyzed (Participants) | 43 | 21 | 48 | 15 | 127
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.7 (8.74) | 68.0 (7.26) | 64.2 (10.72) | 68.7 (8.35) | 65.9 (9.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 6 | 17 | 5 | 38
  Male | 33 | 15 | 31 | 10 | 89
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 40 | 19 | 45 | 13 | 117
  Black | 2 | 2 | 3 | 1 | 8
  Asian | 1 | 0 | 0 | 1 | 2
  American Indian/Alaska native | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Other | 0 | 0 | 0 | 0 | 0
  Multi race | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: Overall response rate is defined as the percentage of participants with an overall response (per the investigator assessment) 2008 Modified International Workshop for Chronic Lymphocytic Leukemia (IWCLL) National Cancer Institute-Working Group (NCI-WG) criteria.
Time Frame: At Wk 5, Day 1; Wk 8, Day 1; Wk 12, Day 1; Wk 16, Day 1; Wk 20, Day 1; Wk 24, Day 1; Wk 36, Day 1; every 12 wks after Wk 36; Final Visit; estimated median time on follow-up was 1694 d for ibrutinib failure cohort and 1942 d for idelalisib failure cohort
Population: All participants in the Main and Expansion Cohorts who received at least one dose of venetoclax
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- ABT-199 After Ibrutinib Therapy: Main and Expansion Cohorts: Participants with ibrutinib-resistant or refractory chronic lymphocytic leukemia (CLL) in the Main and Expansion Cohorts
- ABT-199 After Idelalisib Therapy: Main and Expansion Cohorts: Participants with idelalisib-resistant or refractory chronic lymphocytic leukemia (CLL) in the Main and Expansion Cohorts
Arm/Group | ABT-199 After Ibrutinib Therapy: Main and Expansion Cohorts | ABT-199 After Idelalisib Therapy: Main and Expansion Cohorts
Number analyzed (Participants) | 91 | 36
percentage of participants | 64.8 [54.1 to 74.6] | 69.4 [51.9 to 83.7]

2. Secondary Outcome: Duration of Response (DOR)
Description: DOR is defined as the number of days from the date of first response (complete response [CR], complete response with incomplete marrow recovery [CRi], nodular partial remission [nPR], or partial remission [PR]) to the earliest recurrence or progressive disease. DOR was analyzed by Kaplan-Meier (K-M) methodology.
Time Frame: as for outcome 1
Population: All enrolled participants who received venetoclax, had active disease at baseline, and achieved a response of PR or better
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | ABT-199 After Ibrutinib Therapy: Main and Expansion Cohorts | ABT-199 After Idelalisib Therapy: Main and Expansion Cohorts
Number analyzed (Participants) | 59 | 25
months | 35.1 [19.4 to 50.5] | 55.4 [32.0 to NA] — Not calculable/estimable due to low number of participants with events

3. Secondary Outcome: Time to Progression (TTP)
Description: TTP is defined as the number of days from the date of first dose to the date of earliest disease progression (PD).
  TTP was analyzed by Kaplan-Meier (K-M) methodology.
Time Frame: as for outcome 1
Population: All participants in the Main and Expansion Cohorts who received at least one dose of venetoclax
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | ABT-199 After Ibrutinib Therapy: Main and Expansion Cohorts | ABT-199 After Idelalisib Therapy: Main and Expansion Cohorts
Number analyzed (Participants) | 91 | 36
months | 36.1 [21.9 to 49.0] | 43.4 [20.1 to NA] — Not calculable/estimable due to low number of participants with events

4. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS is defined as the number of days from the date of first dose to the date of earliest disease progression (PD) or death. PFS was analyzed by Kaplan-Meier methodology.
Time Frame: as for outcome 1
Population: All enrolled participants who received venetoclax and had active disease at baseline
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | ABT-199 After Ibrutinib Therapy: Main and Expansion Cohorts | ABT-199 After Idelalisib Therapy: Main and Expansion Cohorts
Number analyzed (Participants) | 91 | 36
months | 24.7 [19.2 to 40.9] | 43.4 [20.1 to NA] — Not calculable/estimable due to low number of participants with events

5. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the number of days from the date of first dose to the date of death for all dosed participants. For participants who did not die, their data was censored at the date of last study visit or the last known date to be alive, whichever was later. OS was estimated using Kaplan-Meier methodology.
Time Frame: as for outcome 1
Population: All participants in the Main and Expansion Cohorts who received at least one dose of venetoclax
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | ABT-199 After Ibrutinib Therapy: Main and Expansion Cohorts | ABT-199 After Idelalisib Therapy: Main and Expansion Cohorts
Number analyzed (Participants) | 91 | 36
months | 69.6 [51.3 to NA] — Not calculable/estimable due to low number of participants with events | NA [57.2 to NA] — Not calculable/estimable due to low number of participants with events

6. Other Pre Specified Outcome: Time to Next Anti-Chronic Lymphocytic Leukemia Treatment (TNNT)
Description: TNNT is defined as the number of days from the date of the first dose of venetoclax to the date of first dose of any non-protocol anti-leukemia therapy (NPT) or death from any cause. For participants who did not take NPT, their data was censored at the last known date to be free of NPT. TTNT was analyzed by Kaplan-Meier methodology.
Time Frame: Collected every 3 months for a period of 5 years after the last participant had enrolled into the study
Population: All participants in the Main and Expansion Cohorts who received at least one dose of venetoclax
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | ABT-199 After Ibrutinib Therapy: Main and Expansion Cohorts | ABT-199 After Idelalisib Therapy: Main and Expansion Cohorts
Number analyzed (Participants) | 91 | 36
months | 24.0 [18.7 to 40.9] | 37.8 [17.1 to NA] — Not calculable/estimable due to low number of participants with events

7. Other Pre Specified Outcome: Percentage of Participants With Minimal Residual Disease (MRD) Negativity Status
Description: The rate of MRD response is defined as the percentage of participants who had MRD negative status.
Time Frame: Assessed at Week 24, Day 1; after the first Complete Response, Complete Remission with Incomplete Marrow Recovery, or Partial Response; at 12-week interval visits until two consecutive negative MRD levels were reported
Population: All participants in the Main and Expansion Cohorts who received at least one dose of venetoclax; indeterminate or missing samples were considered MRD positive for the calculation
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ABT-199 After Ibrutinib Therapy: Main and Expansion Cohorts | ABT-199 After Idelalisib Therapy: Main and Expansion Cohorts
Number analyzed (Participants) | 91 | 36
percentage of participants
  Peripheral blood | 30.8 [21.5 to 41.3] | 25.0 [12.1 to 42.2]
  Bone marrow | 6.6 [2.5 to 13.8] | 11.1 [3.1 to 26.1]

ADVERSE EVENTS:
Time Frame: All-cause mortality reported from enrollment to 30 d after last dose of study drug; median time on follow up was up to 1694 d for those with ibrutinib-resistant or refractory CLL and up to 1942 d for those with idelalisib-resistant or refractory CLL. TEAEs and SAEs collected from first dose of study drug until 30 d after last dose of study drug; mean duration on study drug was 819.8 d (ibrutinib-resistant or refractory CLL cohorts) and 1151.5 d (idelalisib-resistant or refractory CLL cohorts).
Groups:
- ABT-199 After Ibrutinib Therapy: Main Cohort: Participants with ibrutinib-resistant or refractory chronic lymphocytic leukemia (CLL) in the Main Cohort
- ABT-199 After Idelalisib Therapy: Main Cohort: Participants with idelalisib-resistant or refractory chronic lymphocytic leukemia (CLL) in the Main Cohort
- ABT-199 After Ibrutinib or Idelalisib Therapy: Main Cohort: Participants with ibrutinib-resistant/refractory or idelalisib-resistant/refractory chronic lymphocytic leukemia (CLL) in the Main Cohort
- ABT-199 After Ibrutinib Therapy: Expansion Cohort: Participants with ibrutinib-resistant or refractory chronic lymphocytic leukemia (CLL) in the Expansion Cohort
- ABT-199 After Idelalisib Therapy: Expansion Cohort: Participants with idelalisib-resistant or refractory chronic lymphocytic leukemia (CLL) in the Expansion Cohort
- ABT-199 After Ibrutinib or Idelalisib Therapy: Expansion Cohort: Participants with ibrutinib-resistant/refractory or idelalisib-resistant/refractory chronic lymphocytic leukemia (CLL) in the Expansion Cohort
- All Participants: All participants in the Main and Expansion Cohorts
Arm/Group | ABT-199 After Ibrutinib Therapy: Main Cohort | ABT-199 After Idelalisib Therapy: Main Cohort | ABT-199 After Ibrutinib or Idelalisib Therapy: Main Cohort | ABT-199 After Ibrutinib Therapy: Expansion Cohort | ABT-199 After Idelalisib Therapy: Expansion Cohort | ABT-199 After Ibrutinib or Idelalisib Therapy: Expansion Cohort | ABT-199 After Ibrutinib Therapy: Main and Expansion Cohorts | ABT-199 After Idelalisib Therapy: Main and Expansion Cohorts | All Participants
All-Cause Mortality (participants affected / at risk) | 25/43 | 9/21 | 34/64 | 17/48 | 4/15 | 21/63 | 42/91 | 13/36 | 55/127
Serious Adverse Events (participants affected / at risk) | 35/43 | 14/21 | 49/64 | 26/48 | 9/15 | 35/63 | 61/91 | 23/36 | 84/127
Other Adverse Events (participants affected / at risk) | 43/43 | 21/21 | 64/64 | 48/48 | 15/15 | 63/63 | 91/91 | 36/36 | 127/127
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ABT-199 After Ibrutinib Therapy: Main Cohort (N=43) | ABT-199 After Idelalisib Therapy: Main Cohort (N=21) | ABT-199 After Ibrutinib or Idelalisib Therapy: Main Cohort (N=64) | ABT-199 After Ibrutinib Therapy: Expansion Cohort (N=48) | ABT-199 After Idelalisib Therapy: Expansion Cohort (N=15) | ABT-199 After Ibrutinib or Idelalisib Therapy: Expansion Cohort (N=63) | ABT-199 After Ibrutinib Therapy: Main and Expansion Cohorts (N=91) | ABT-199 After Idelalisib Therapy: Main and Expansion Cohorts (N=36) | All Participants (N=127)
ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 2 (2)
AUTOIMMUNE HAEMOLYTIC ANAEMIA (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 2 (3)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 10 (13) | 1 (1) | 11 (14) | 3 (4) | 0 (0) | 3 (4) | 13 (17) | 1 (1) | 14 (18)
HAEMOLYTIC ANAEMIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
LYMPHOPENIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
NEUTROPENIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
ANGINA UNSTABLE (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
ATRIAL FIBRILLATION (Cardiac disorders) | 0 (0) | 1 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2)
ATRIAL FLUTTER (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
MYOCARDIAL INFARCTION (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 2 (2)
VENTRICULAR TACHYCARDIA (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
DIARRHOEA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
DYSPEPSIA (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
DYSPHAGIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
EROSIVE OESOPHAGITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
GASTRIC ULCER (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
INCARCERATED INGUINAL HERNIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
INTESTINAL ISCHAEMIA (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
MESENTERIC VEIN THROMBOSIS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
MOUTH HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 1 (2) | 2 (3) | 0 (0) | 2 (3)
STOMATITIS (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
ASTHENIA (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
CHEST PAIN (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 2 (2)
DEATH (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
DISEASE PROGRESSION (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 2 (2)
FACIAL PAIN (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
FATIGUE (General disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
MULTIPLE ORGAN DYSFUNCTION SYNDROME (General disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 3 (3)
PYREXIA (General disorders) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 1 (1) | 3 (3) | 2 (2) | 3 (3) | 5 (5)
SYSTEMIC INFLAMMATORY RESPONSE SYNDROME (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
BILE DUCT STONE (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
CYTOKINE RELEASE SYNDROME (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 2 (2)
APPENDICITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
ARTHRITIS BACTERIAL (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
BACTERAEMIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 3 (3) | 3 (3) | 0 (0) | 3 (3)
BRONCHITIS (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
CELLULITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 2 (3) | 2 (3) | 0 (0) | 2 (3)
CORYNEBACTERIUM BACTERAEMIA (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
CORYNEBACTERIUM SEPSIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
DIVERTICULITIS (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
ESCHERICHIA BACTERAEMIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
ESCHERICHIA SEPSIS (Infections and infestations) | 1 (2) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (2)
GASTROENTERITIS (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
GASTROENTERITIS VIRAL (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
INFLUENZA (Infections and infestations) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
LYMPH GLAND INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
PAROTITIS (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
PHARYNGITIS (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
PNEUMONIA (Infections and infestations) | 6 (8) | 3 (8) | 9 (16) | 3 (4) | 1 (1) | 4 (5) | 9 (12) | 4 (9) | 13 (21)
PNEUMONIA ASPIRATION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
PNEUMONIA BACTERIAL (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
PNEUMONIA LEGIONELLA (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
PNEUMONIA PSEUDOMONAL (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (2) | 1 (2) | 0 (0) | 1 (2)
PNEUMONIA VIRAL (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
RHINOVIRUS INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 2 (2)
SEPSIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 3 (3) | 1 (1) | 2 (2) | 3 (3)
SEPTIC SHOCK (Infections and infestations) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
STAPHYLOCOCCAL BACTERAEMIA (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
STREPTOCOCCAL BACTERAEMIA (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
WOUND INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
FALL (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
JOINT DISLOCATION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
PELVIC FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
POST PROCEDURAL HAEMATURIA (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
BLOOD CREATININE INCREASED (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
BLOOD GLUCOSE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
BLOOD POTASSIUM INCREASED (Investigations) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 3 (3)
DEHYDRATION (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 2 (2)
HYPERCALCAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 4 (4) | 4 (4) | 1 (1) | 5 (5)
HYPERKALAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
HYPERPHOSPHATAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
HYPERVOLAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
GROIN PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
LUMBAR SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
ADENOCARCINOMA OF COLON (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 2 (2)
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
BLADDER CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
CHRONIC LYMPHOCYTIC LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
HIGH-GRADE B-CELL LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
MALIGNANT NEOPLASM PROGRESSION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
METASTASES TO MENINGES (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
MUCOEPIDERMOID CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
MYELODYSPLASTIC SYNDROME (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
RICHTER'S SYNDROME (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
SALIVARY GLAND CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
CAUDA EQUINA SYNDROME (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
HAEMORRHAGE INTRACRANIAL (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
PARAESTHESIA (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
PRESYNCOPE (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 2 (2)
SEIZURE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
BLADDER OUTLET OBSTRUCTION (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
NEPHROLITHIASIS (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
RENAL FAILURE (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
URINARY TRACT OBSTRUCTION (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
BENIGN PROSTATIC HYPERPLASIA (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
PROSTATIC OBSTRUCTION (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
ASPHYXIA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 2 (2)
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
PULMONARY GRANULOMA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 2 (2)
DRUG ERUPTION (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
EOSINOPHILIC CELLULITIS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
ORTHOSTATIC HYPOTENSION (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ABT-199 After Ibrutinib Therapy: Main Cohort (N=43) | ABT-199 After Idelalisib Therapy: Main Cohort (N=21) | ABT-199 After Ibrutinib or Idelalisib Therapy: Main Cohort (N=64) | ABT-199 After Ibrutinib Therapy: Expansion Cohort (N=48) | ABT-199 After Idelalisib Therapy: Expansion Cohort (N=15) | ABT-199 After Ibrutinib or Idelalisib Therapy: Expansion Cohort (N=63) | ABT-199 After Ibrutinib Therapy: Main and Expansion Cohorts (N=91) | ABT-199 After Idelalisib Therapy: Main and Expansion Cohorts (N=36) | All Participants (N=127)
ANAEMIA (Blood and lymphatic system disorders) | 24 (44) | 4 (25) | 28 (69) | 21 (51) | 3 (3) | 24 (54) | 45 (95) | 7 (28) | 52 (123)
LYMPH NODE PAIN (Blood and lymphatic system disorders) | 3 (3) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 4 (4)
NEUTROPENIA (Blood and lymphatic system disorders) | 16 (32) | 10 (27) | 26 (59) | 20 (44) | 9 (15) | 29 (59) | 36 (76) | 19 (42) | 55 (118)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 11 (14) | 6 (24) | 17 (38) | 14 (25) | 4 (7) | 18 (32) | 25 (39) | 10 (31) | 35 (70)
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 3 (3) | 1 (1) | 4 (4) | 1 (1) | 1 (1) | 2 (2) | 4 (4) | 2 (2) | 6 (6)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 3 (3) | 0 (0) | 3 (3) | 5 (5) | 2 (2) | 7 (7) | 8 (8) | 2 (2) | 10 (10)
ABDOMINAL PAIN (Gastrointestinal disorders) | 7 (10) | 0 (0) | 7 (10) | 13 (16) | 3 (5) | 16 (21) | 20 (26) | 3 (5) | 23 (31)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1 (2) | 1 (1) | 2 (3) | 3 (3) | 3 (4) | 6 (7) | 4 (5) | 4 (5) | 8 (10)
CONSTIPATION (Gastrointestinal disorders) | 7 (12) | 7 (7) | 14 (19) | 17 (18) | 3 (4) | 20 (22) | 24 (30) | 10 (11) | 34 (41)
DIARRHOEA (Gastrointestinal disorders) | 22 (38) | 9 (18) | 31 (56) | 26 (56) | 8 (15) | 34 (71) | 48 (94) | 17 (33) | 65 (127)
DRY MOUTH (Gastrointestinal disorders) | 2 (2) | 3 (3) | 5 (5) | 5 (5) | 0 (0) | 5 (5) | 7 (7) | 3 (3) | 10 (10)
DYSPEPSIA (Gastrointestinal disorders) | 3 (3) | 1 (2) | 4 (5) | 1 (1) | 0 (0) | 1 (1) | 4 (4) | 1 (2) | 5 (6)
DYSPHAGIA (Gastrointestinal disorders) | 3 (3) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 4 (4) | 0 (0) | 4 (4)
FLATULENCE (Gastrointestinal disorders) | 3 (3) | 1 (1) | 4 (4) | 3 (3) | 1 (1) | 4 (4) | 6 (6) | 2 (2) | 8 (8)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 4 (4) | 3 (3) | 7 (7) | 5 (5) | 1 (1) | 6 (6) | 9 (9) | 4 (4) | 13 (13)
HAEMORRHOIDS (Gastrointestinal disorders) | 4 (4) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 4 (4)
LARGE INTESTINE POLYP (Gastrointestinal disorders) | 1 (1) | 2 (3) | 3 (4) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 2 (3) | 4 (5)
NAUSEA (Gastrointestinal disorders) | 24 (32) | 6 (9) | 30 (41) | 30 (38) | 4 (8) | 34 (46) | 54 (70) | 10 (17) | 64 (87)
ORAL PAIN (Gastrointestinal disorders) | 3 (3) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 2 (2) | 4 (4) | 1 (1) | 5 (5)
STOMATITIS (Gastrointestinal disorders) | 4 (4) | 0 (0) | 4 (4) | 5 (5) | 1 (1) | 6 (6) | 9 (9) | 1 (1) | 10 (10)
TOOTHACHE (Gastrointestinal disorders) | 3 (3) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 3 (3)
VOMITING (Gastrointestinal disorders) | 10 (18) | 3 (9) | 13 (27) | 16 (27) | 0 (0) | 16 (27) | 26 (45) | 3 (9) | 29 (54)
CHILLS (General disorders) | 4 (4) | 3 (4) | 7 (8) | 8 (9) | 0 (0) | 8 (9) | 12 (13) | 3 (4) | 15 (17)
FATIGUE (General disorders) | 20 (28) | 7 (9) | 27 (37) | 22 (31) | 3 (6) | 25 (37) | 42 (59) | 10 (15) | 52 (74)
INFLUENZA LIKE ILLNESS (General disorders) | 1 (2) | 3 (3) | 4 (5) | 5 (5) | 0 (0) | 5 (5) | 6 (7) | 3 (3) | 9 (10)
NON-CARDIAC CHEST PAIN (General disorders) | 0 (0) | 1 (1) | 1 (1) | 4 (4) | 0 (0) | 4 (4) | 4 (4) | 1 (1) | 5 (5)
OEDEMA (General disorders) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 3 (3)
OEDEMA PERIPHERAL (General disorders) | 8 (8) | 6 (8) | 14 (16) | 18 (19) | 1 (2) | 19 (21) | 26 (27) | 7 (10) | 33 (37)
PAIN (General disorders) | 3 (3) | 1 (1) | 4 (4) | 3 (3) | 1 (1) | 4 (4) | 6 (6) | 2 (2) | 8 (8)
PERIPHERAL SWELLING (General disorders) | 1 (1) | 3 (3) | 4 (4) | 2 (2) | 1 (1) | 3 (3) | 3 (3) | 4 (4) | 7 (7)
PYREXIA (General disorders) | 5 (6) | 3 (3) | 8 (9) | 11 (18) | 2 (2) | 13 (20) | 16 (24) | 5 (5) | 21 (29)
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 5 (5) | 4 (4) | 1 (1) | 5 (5)
SEASONAL ALLERGY (Immune system disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
BRONCHITIS (Infections and infestations) | 2 (2) | 1 (1) | 3 (3) | 4 (5) | 3 (4) | 7 (9) | 6 (7) | 4 (5) | 10 (12)
CELLULITIS (Infections and infestations) | 2 (2) | 3 (4) | 5 (6) | 3 (4) | 0 (0) | 3 (4) | 5 (6) | 3 (4) | 8 (10)
CONJUNCTIVITIS (Infections and infestations) | 1 (1) | 2 (2) | 3 (3) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 3 (3) | 5 (5)
HERPES ZOSTER (Infections and infestations) | 1 (1) | 2 (3) | 3 (4) | 2 (2) | 0 (0) | 2 (2) | 3 (3) | 2 (3) | 5 (6)
INFLUENZA (Infections and infestations) | 5 (5) | 3 (4) | 8 (9) | 3 (3) | 1 (1) | 4 (4) | 8 (8) | 4 (5) | 12 (13)
NASOPHARYNGITIS (Infections and infestations) | 5 (5) | 1 (1) | 6 (6) | 2 (2) | 1 (2) | 3 (4) | 7 (7) | 2 (3) | 9 (10)
ORAL CANDIDIASIS (Infections and infestations) | 1 (1) | 2 (2) | 3 (3) | 1 (2) | 0 (0) | 1 (2) | 2 (3) | 2 (2) | 4 (5)
PNEUMONIA (Infections and infestations) | 4 (4) | 3 (3) | 7 (7) | 2 (2) | 1 (1) | 3 (3) | 6 (6) | 4 (4) | 10 (10)
SINUSITIS (Infections and infestations) | 2 (2) | 1 (1) | 3 (3) | 6 (7) | 3 (5) | 9 (12) | 8 (9) | 4 (6) | 12 (15)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 15 (29) | 9 (15) | 24 (44) | 19 (37) | 7 (16) | 26 (53) | 34 (66) | 16 (31) | 50 (97)
URINARY TRACT INFECTION (Infections and infestations) | 2 (5) | 2 (8) | 4 (13) | 9 (17) | 0 (0) | 9 (17) | 11 (22) | 2 (8) | 13 (30)
CONTUSION (Injury, poisoning and procedural complications) | 10 (11) | 2 (2) | 12 (13) | 9 (10) | 1 (1) | 10 (11) | 19 (21) | 3 (3) | 22 (24)
FALL (Injury, poisoning and procedural complications) | 3 (3) | 1 (1) | 4 (4) | 4 (6) | 1 (1) | 5 (7) | 7 (9) | 2 (2) | 9 (11)
SKIN ABRASION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 4 (5) | 0 (0) | 4 (5) | 5 (6) | 0 (0) | 5 (6)
SKIN LACERATION (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 4 (4) | 2 (2) | 1 (1) | 3 (3) | 4 (4) | 3 (3) | 7 (7)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 6 (8) | 2 (7) | 8 (15) | 8 (8) | 0 (0) | 8 (8) | 14 (16) | 2 (7) | 16 (23)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 10 (13) | 2 (3) | 12 (16) | 8 (9) | 2 (6) | 10 (15) | 18 (22) | 4 (9) | 22 (31)
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 4 (4) | 2 (4) | 6 (8) | 5 (5) | 2 (4) | 7 (9) | 9 (9) | 4 (8) | 13 (17)
BLOOD BILIRUBIN INCREASED (Investigations) | 4 (4) | 3 (3) | 7 (7) | 8 (12) | 2 (2) | 10 (14) | 12 (16) | 5 (5) | 17 (21)
BLOOD CHOLESTEROL INCREASED (Investigations) | 0 (0) | 2 (2) | 2 (2) | 2 (3) | 0 (0) | 2 (3) | 2 (3) | 2 (2) | 4 (5)
BLOOD CREATININE INCREASED (Investigations) | 2 (3) | 2 (3) | 4 (6) | 6 (10) | 3 (7) | 9 (17) | 8 (13) | 5 (10) | 13 (23)
LYMPHOCYTE COUNT DECREASED (Investigations) | 12 (28) | 2 (2) | 14 (30) | 12 (27) | 1 (1) | 13 (28) | 24 (55) | 3 (3) | 27 (58)
LYMPHOCYTE COUNT INCREASED (Investigations) | 6 (10) | 0 (0) | 6 (10) | 2 (2) | 0 (0) | 2 (2) | 8 (12) | 0 (0) | 8 (12)
NEUTROPHIL COUNT DECREASED (Investigations) | 20 (60) | 1 (1) | 21 (61) | 12 (48) | 2 (2) | 14 (50) | 32 (108) | 3 (3) | 35 (111)
PLATELET COUNT DECREASED (Investigations) | 19 (35) | 1 (1) | 20 (36) | 11 (23) | 4 (6) | 15 (29) | 30 (58) | 5 (7) | 35 (65)
WEIGHT DECREASED (Investigations) | 4 (6) | 1 (1) | 5 (7) | 6 (6) | 0 (0) | 6 (6) | 10 (12) | 1 (1) | 11 (13)
WEIGHT INCREASED (Investigations) | 3 (3) | 1 (1) | 4 (4) | 5 (7) | 1 (1) | 6 (8) | 8 (10) | 2 (2) | 10 (12)
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 18 (40) | 2 (6) | 20 (46) | 16 (64) | 3 (4) | 19 (68) | 34 (104) | 5 (10) | 39 (114)
DECREASED APPETITE (Metabolism and nutrition disorders) | 5 (5) | 3 (3) | 8 (8) | 3 (3) | 3 (3) | 6 (6) | 8 (8) | 6 (6) | 14 (14)
DEHYDRATION (Metabolism and nutrition disorders) | 5 (6) | 2 (2) | 7 (8) | 2 (2) | 1 (1) | 3 (3) | 7 (8) | 3 (3) | 10 (11)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 3 (4) | 3 (8) | 6 (12) | 7 (18) | 0 (0) | 7 (18) | 10 (22) | 3 (8) | 13 (30)
HYPERKALAEMIA (Metabolism and nutrition disorders) | 7 (9) | 1 (2) | 8 (11) | 6 (11) | 2 (3) | 8 (14) | 13 (20) | 3 (5) | 16 (25)
HYPERNATRAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 0 (0) | 4 (5) | 4 (5) | 0 (0) | 4 (5)
HYPERPHOSPHATAEMIA (Metabolism and nutrition disorders) | 7 (9) | 6 (8) | 13 (17) | 4 (7) | 1 (1) | 5 (8) | 11 (16) | 7 (9) | 18 (25)
HYPERURICAEMIA (Metabolism and nutrition disorders) | 10 (22) | 4 (7) | 14 (29) | 4 (5) | 2 (6) | 6 (11) | 14 (27) | 6 (13) | 20 (40)
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 6 (10) | 1 (3) | 7 (13) | 10 (20) | 2 (6) | 12 (26) | 16 (30) | 3 (9) | 19 (39)
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 9 (17) | 3 (6) | 12 (23) | 14 (28) | 3 (5) | 17 (33) | 23 (45) | 6 (11) | 29 (56)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 11 (15) | 5 (11) | 16 (26) | 13 (25) | 4 (9) | 17 (34) | 24 (40) | 9 (20) | 33 (60)
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 10 (17) | 1 (1) | 11 (18) | 14 (16) | 3 (4) | 17 (20) | 24 (33) | 4 (5) | 28 (38)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 12 (16) | 2 (3) | 14 (19) | 7 (12) | 2 (4) | 9 (16) | 19 (28) | 4 (7) | 23 (35)
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 6 (10) | 3 (3) | 9 (13) | 12 (17) | 4 (7) | 16 (24) | 18 (27) | 7 (10) | 25 (37)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 5 (7) | 3 (3) | 8 (10) | 15 (31) | 3 (5) | 18 (36) | 20 (38) | 6 (8) | 26 (46)
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 3 (4) | 0 (0) | 3 (4) | 2 (2) | 1 (1) | 3 (3) | 5 (6) | 1 (1) | 6 (7)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 8 (8) | 4 (4) | 12 (12) | 10 (16) | 3 (3) | 13 (19) | 18 (24) | 7 (7) | 25 (31)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 3 (4) | 0 (0) | 3 (4) | 2 (2) | 1 (1) | 3 (3) | 5 (6) | 1 (1) | 6 (7)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 5 (5) | 5 (5) | 10 (10) | 4 (5) | 1 (1) | 5 (6) | 9 (10) | 6 (6) | 15 (16)
MUSCLE TIGHTNESS (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 3 (3)
MYALGIA (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (4) | 5 (8) | 3 (3) | 1 (1) | 4 (4) | 7 (7) | 2 (5) | 9 (12)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 6 (6) | 4 (5) | 10 (11) | 9 (11) | 4 (4) | 13 (15) | 15 (17) | 8 (9) | 23 (26)
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 2 (2) | 5 (5) | 4 (5) | 2 (2) | 6 (7) | 7 (8) | 4 (4) | 11 (12)
SQUAMOUS CELL CARCINOMA OF SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (5) | 1 (1) | 3 (6) | 4 (6) | 2 (2) | 6 (8) | 6 (11) | 3 (3) | 9 (14)
DIZZINESS (Nervous system disorders) | 6 (8) | 1 (1) | 7 (9) | 13 (14) | 4 (4) | 17 (18) | 19 (22) | 5 (5) | 24 (27)
HEADACHE (Nervous system disorders) | 12 (14) | 4 (6) | 16 (20) | 15 (24) | 2 (2) | 17 (26) | 27 (38) | 6 (8) | 33 (46)
HYPOAESTHESIA (Nervous system disorders) | 3 (3) | 0 (0) | 3 (3) | 3 (3) | 1 (1) | 4 (4) | 6 (6) | 1 (1) | 7 (7)
PARAESTHESIA (Nervous system disorders) | 2 (2) | 2 (3) | 4 (5) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 3 (4) | 5 (6)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 4 (5) | 1 (1) | 5 (6) | 5 (6) | 1 (1) | 6 (7)
ANXIETY (Psychiatric disorders) | 1 (1) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 3 (3)
DEPRESSION (Psychiatric disorders) | 1 (1) | 2 (3) | 3 (4) | 3 (3) | 2 (2) | 5 (5) | 4 (4) | 4 (5) | 8 (9)
INSOMNIA (Psychiatric disorders) | 3 (5) | 6 (6) | 9 (11) | 10 (10) | 2 (2) | 12 (12) | 13 (15) | 8 (8) | 21 (23)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 4 (4) | 2 (2) | 6 (6) | 2 (2) | 1 (1) | 3 (3) | 6 (6) | 3 (3) | 9 (9)
BLADDER SPASM (Renal and urinary disorders) | 1 (1) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 3 (3)
POLLAKIURIA (Renal and urinary disorders) | 2 (2) | 3 (3) | 5 (5) | 3 (3) | 1 (1) | 4 (4) | 5 (5) | 4 (4) | 9 (9)
ERECTILE DYSFUNCTION (Reproductive system and breast disorders) | 3 (3) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 3 (3)
COUGH (Respiratory, thoracic and mediastinal disorders) | 14 (18) | 4 (5) | 18 (23) | 13 (17) | 5 (7) | 18 (24) | 27 (35) | 9 (12) | 36 (47)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 13 (17) | 3 (3) | 16 (20) | 7 (9) | 3 (3) | 10 (12) | 20 (26) | 6 (6) | 26 (32)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 0 (0) | 4 (5) | 6 (7) | 0 (0) | 6 (7) | 10 (12) | 0 (0) | 10 (12)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 4 (5) | 10 (12) | 2 (2) | 1 (1) | 3 (3) | 8 (9) | 5 (6) | 13 (15)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 1 (1) | 7 (7) | 7 (10) | 1 (1) | 8 (11) | 13 (16) | 2 (2) | 15 (18)
RHINITIS ALLERGIC (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 3 (3) | 4 (6) | 1 (1) | 5 (7) | 7 (9) | 1 (1) | 8 (10)
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4) | 5 (5) | 2 (4) | 2 (2) | 4 (6) | 3 (5) | 6 (6) | 9 (11)
SINUS CONGESTION (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 0 (0) | 3 (4) | 0 (0) | 1 (1) | 1 (1) | 3 (4) | 1 (1) | 4 (5)
UPPER-AIRWAY COUGH SYNDROME (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 2 (2) | 5 (7) | 6 (6) | 0 (0) | 6 (6) | 9 (11) | 2 (2) | 11 (13)
WHEEZING (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 2 (2) | 4 (6) | 2 (2) | 0 (0) | 2 (2) | 4 (6) | 2 (2) | 6 (8)
ACTINIC KERATOSIS (Skin and subcutaneous tissue disorders) | 4 (5) | 2 (2) | 6 (7) | 1 (1) | 0 (0) | 1 (1) | 5 (6) | 2 (2) | 7 (8)
DRY SKIN (Skin and subcutaneous tissue disorders) | 3 (5) | 0 (0) | 3 (5) | 3 (4) | 0 (0) | 3 (4) | 6 (9) | 0 (0) | 6 (9)
ECZEMA (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 3 (3) | 2 (2) | 0 (0) | 2 (2) | 3 (3) | 2 (2) | 5 (5)
HAIR COLOUR CHANGES (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 3 (3)
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 4 (4) | 1 (1) | 5 (5) | 3 (3) | 0 (0) | 3 (3) | 7 (7) | 1 (1) | 8 (8)
NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 5 (6) | 0 (0) | 5 (6) | 6 (6) | 0 (0) | 6 (6) | 11 (12) | 0 (0) | 11 (12)
PRURITUS (Skin and subcutaneous tissue disorders) | 4 (5) | 4 (6) | 8 (11) | 1 (1) | 2 (2) | 3 (3) | 5 (6) | 6 (8) | 11 (14)
RASH (Skin and subcutaneous tissue disorders) | 8 (8) | 6 (12) | 14 (20) | 6 (7) | 3 (4) | 9 (11) | 14 (15) | 9 (16) | 23 (31)
SKIN LESION (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 2 (2) | 5 (5) | 0 (0) | 5 (5)
SKIN ULCER (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 2 (2) | 5 (5) | 0 (0) | 5 (5)
HYPERTENSION (Vascular disorders) | 7 (12) | 3 (3) | 10 (15) | 11 (15) | 4 (7) | 15 (22) | 18 (27) | 7 (10) | 25 (37)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2020-12-15): https://cdn.clinicaltrials.gov/large-docs/82/NCT02141282/Prot_000.pdf
  • Statistical Analysis Plan (2018-11-09): https://cdn.clinicaltrials.gov/large-docs/82/NCT02141282/SAP_001.pdf